CLINICAL TRIAL: NCT06020963
Title: Can Acupoint Low Intensity Shockwave Therapy Improve Bladder Voiding Efficiency: A Pilot Study.
Brief Title: Can Acupoint Low Intensity Shockwave Therapy Improve Bladder Voiding Efficiency
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Armed Forces General Hospital (Other Government)
Responsible Party: Principal Investigator, Jing-Dung, SHEN, Director of Urology, Taichung Armed Forces General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A202205205
Record Dates: First submitted 2023-08-27; First posted 2023-09-01 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Detrusor Underactivity
Keywords: detrusor underactivity; acupoint; voiding dysfunction; bladder voiding efficiency; low-intensity extracorporeal shockwave therapy
MeSH Terms: conditions — Urinary Bladder, Underactive | interventions — Tamsulosin

STUDY DESIGN:
Intervention Model Description: Evaluate the treatment effect of Low-intensity shockwave therapy on acupoint (CV-4, ST-28, SP-6 once a week for 8 weeks) and the control group is oral tamsulosin 0.2mg daily for 8 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group-1 (Experimental): Low intensive shockwave therapy 1000 shocks on each acupoint (CV-4, and bilateral ST-28) once a week for 8 weeks.
  Interventions: Procedure: Low Intensity Shockwave Therapy (LiSWT)
- Group-2 (Experimental): Low intensive shockwave therapy 1000 shocks on each acupoint (CV-4, and bilateral SP-6) once a week for 8 weeks.
  Interventions: Procedure: Low Intensity Shockwave Therapy (LiSWT)
- Group-3 (Active Comparator): Oral tamsulosin 0.2mg once daily for 8 weeks.
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Procedure: Low Intensity Shockwave Therapy (LiSWT) — Low Intensity Shockwave Therapy (LiSWT) has been used for many years. Its mechanism is to use shock wave energy to promote angiogenesis to achieve the functions of tissue repair and cell regeneration.
  Arms: Group-1; Group-2
Drug: Tamsulosin — Tamsulosin is a selective alpha-1 blocker, its main function is to relax the smooth muscles of the base of the prostate, urethra, and bladder, and improve lower urinary tract symptoms.
  Other Names: Harnalidge 0.2mg
  Arms: Group-3

SUMMARY:
With the increasing of the elderly population, patients with urinary dysfunction caused by inefficiency of bladder emptying becomes much often than before. However, the current treatments for this kind of bladder dysfunction are limited and unsatisfactory. Low-intensity extracorporeal shockwave therapy (LiESWT) is a very popular emerging treatment in recent years, and abundant of literatures have confirmed that this treatment is safe and effective in myofascial pain and male erectile dysfunction. Recently, many animal experiments have showed that LiESWT could improve urinary dysfunction caused by bladder dysfunction. Taiwan based studies also reported that LiESWT could improve symptoms of overactive bladder. LiESWT is a non-drug, low-invasive and high-safety treatment, which is very suitable for elderly patients. In this study investigator combine the LiESWT and acupuncture to treat the patients with underactive bladder. Investigator hypothesize that LiESWT could improve bladder voiding efficiency.

DETAILED DESCRIPTION:
This is a randomized controlled trial, the inclusion criteria are the patients more than 20 years old and bladder voiding efficiency less than 70%, this trial will enroll 60 male and 40 female , total 100 patients. The male will be randomly assigned into three groups(Group-1, Group-2, Group-3) by ratio 1:1:1, and the female will be randomly assigned into two groups (Group-1, Group-2) by ratio 1:1. Group-1: LiESWT on acupoint CV-4, and bilateral ST-28 once a week for 8 weeks, Group-2: LiESWT on acupoint CV-4 and bilateral acupoint SP-6 once a week for 8 weeks, Group-3: Treatment with oral tamsulosin 0.2mg per-day for 8 weeks. The primary outcome is the improvement of bladder voiding efficiency. The secondary outcomes are global response assessment scale, the improvement of maximum uroflow rate, post-voiding residual urine amount, total score of international prostate symptom score.

ELIGIBILITY:
Inclusion Criteria:

1.Bladder voiding efficiency is less than 70%.

Exclusion Criteria:

1. Patient who has history active pelvic malignancy without treatment.
2. Acute urinary tract infection.
3. Pregnancy
4. Active infective lesion on treatment site.
5. Open wound on treatment site.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Bladder Voiding Efficiency (BVE) | Baseline, Week 4, Week 8, Week 12
  Bladder Voiding Efficiency (BVE) is the ratio of the voiding volume of urine over total bladder urine volume

SECONDARY OUTCOMES:
Global Response Assessment scale | Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 12.
  GRA is a scale for subjective evaluation of treatment effects by patients, ranging from the worst -3 points to the best 3 points
Maximum uroflow rate | Baseline, Week 4, Week 8, Week 12
  The maximum uroflow rate during voiding.
Post-Voiding Residual urine amount | Baseline, Week 4, Week 8, Week 12
  Post-Voiding Residual urine amount is the residual urine in bladder after voiding.
Total score of international prostate symptom score | Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 12.
  International prostate symptom score is a questionnaire used to assess the severity of lower urinary tract symptoms, ranging from best 0, to the worst 35.

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Dung Shen, MD, Principal Investigator — Taichung Armed Forces General Hospital
Locations (1):
- Taichung Armed Forces General Hospital, Taichung, Other (Non US), Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simplicio CL, Purita J, Murrell W, Santos GS, Dos Santos RG, Lana JFSD. Extracorporeal shock wave therapy mechanisms in musculoskeletal regenerative medicine. J Clin Orthop Trauma. 2020 May;11(Suppl 3):S309-S318. doi: 10.1016/j.jcot.2020.02.004. Epub 2020 Feb 12. PMID 32523286
- [Background] Lee YC, Hsieh TJ, Tang FH, Jhan JH, Lin KL, Juan YS, Wang HS, Long CY. Therapeutic effect of Low intensity Extracorporeal Shock Wave Therapy (Li-ESWT) on diabetic bladder dysfunction in a rat model. Int J Med Sci. 2021 Jan 29;18(6):1423-1431. doi: 10.7150/ijms.55274. eCollection 2021. PMID 33628099
- [Background] Wang HS, Oh BS, Wang B, Ruan Y, Zhou J, Banie L, Lee YC, Tamaddon A, Zhou T, Wang G, Lin G, Lue TF. Low-intensity extracorporeal shockwave therapy ameliorates diabetic underactive bladder in streptozotocin-induced diabetic rats. BJU Int. 2018 Sep;122(3):490-500. doi: 10.1111/bju.14216. Epub 2018 Apr 20. PMID 29603534
- [Background] Dimitriadis F, Papaioannou M, Sokolakis I, Fragou A, Hatzichristou D, Apostolidis A. The Effect of Low-Intensity Extracorporeal Shockwave Treatment on the Urinary Bladder in an Experimental Diabetic Rat Model. Int Neurourol J. 2021 Mar;25(1):34-41. doi: 10.5213/inj.2040344.172. Epub 2021 Mar 6. PMID 33676379
- [Background] Chuang YC, Tyagi P, Luo HL, Lee WC, Wang HJ, Huang CC, Chancellor MB. Long-term functional change of cryoinjury-induced detrusor underactivity and effects of extracorporeal shock wave therapy in a rat model. Int Urol Nephrol. 2019 Apr;51(4):617-626. doi: 10.1007/s11255-019-02095-4. Epub 2019 Feb 22. PMID 30796726
- [Background] Chuang YC, Tyagi P, Wang HJ, Huang CC, Lin CC, Chancellor MB. Urodynamic and molecular characteristics of detrusor underactivity in a rat cryoinjury model and effects of low energy shock wave therapy. Neurourol Urodyn. 2018 Feb;37(2):708-715. doi: 10.1002/nau.23381. Epub 2017 Aug 2. PMID 28767169
- [Background] Yoshida M, Sekido N, Matsukawa Y, Yono M, Yamaguchi O. Clinical diagnostic criteria for detrusor underactivity: A report from the Japanese Continence Society working group on underactive bladder. Low Urin Tract Symptoms. 2021 Jan;13(1):13-16. doi: 10.1111/luts.12356. Epub 2020 Oct 7. PMID 33029933
- [Background] Lin KL, Lu JH, Chueh KS, Juan TJ, Wu BN, Chuang SM, Lee YC, Shen MC, Long CY, Juan YS. Low-Intensity Extracorporeal Shock Wave Therapy Promotes Bladder Regeneration and Improves Overactive Bladder Induced by Ovarian Hormone Deficiency from Rat Animal Model to Human Clinical Trial. Int J Mol Sci. 2021 Aug 27;22(17):9296. doi: 10.3390/ijms22179296. PMID 34502202